CLINICAL TRIAL: NCT02331797
Title: Endoscopic Overlay Tympanoplasty in Correcting Large Tympanic Membrane Perforation
Brief Title: Endoscopic Overlay Tympanoplasty for TM Perforation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Yuvatiya Plodpai, Doctor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 57-0123-13-1
Record Dates: First submitted 2014-12-26; First posted 2015-01-06 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Tympanic Membrane Perforation
Keywords: endoscope; microscope; transcanal
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic Technique (Experimental): All patients are operated under the endoscope. The endoscope passed through external auditory canal (transcanal approach) to visualize tympanic remnant.
  Interventions: Device: Endoscopic Technique
- Microscopic Technique (Active Comparator): All patients are operated under the microscope.A postauricular or transcanal approach is chose depend on ear canal size and size of perforation. When the ear canal is too small, the postauricular is used.
  Interventions: Device: Microscopic Technique

INTERVENTIONS:
Device: Endoscopic Technique — Endoscopic Technique; endoscopic transcanal lateral graft tympanoplasty using An endoscope (Karl Storz, Tuttlingen, Germany) and A microdrill (Skeeter Otologic Drill System; Medtronic Xom ed Surgical Products, Inc., Jacksonville, FL, USA)
  Arms: Endoscopic Technique
Device: Microscopic Technique — Microsopic surgical approach using a Zeiss Opmi 111 (Carl Zeiss, Jena, Germany) operating microscope
  Arms: Microscopic Technique

SUMMARY:
Minimally invasive surgery is becoming more common in many surgical fields. The wide view of endoscope allows for minimally invasive transcanal approach instead of large postauricular opening. The investigators conduct this study to compared post operative pain score (by Visual Analogue Scales) between conventional microscope lateral placing tympanoplasty and endoscopic lateral placing tympanoplasty.

DETAILED DESCRIPTION:
A main part of tympanoplasty is repair of perforated tympanic membrane. There are two popular way to approach tympanic membrane, transcanal or postauricular approach. There are two grafting techniques are applied in tympanoplasty which includes the lateral technique (overlay) and medial technique (underlay).

The lateral technique is widely used in our institute which involves placement of a graft lateral to the tympanic annulus and the fibrous layer of the tympanic remnant. The most our preferred approach in previous experience is the postauricular approach for tympanoplasty because the transcanal approach is not enough for adequate exposure. Moreover, the visualization straight through transcanal provide by the microscope is difficult by a limited view of the perforation edge due to narrowing and curved external ear canal. Postauricular approach cause many layers of tissue are violated along with a significant postoperative pain.

The author proposed this study with the aim of determining the alleviation of postoperative pain by new technique and the efficacy of endoscope for tympanoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-70 years
* The patients who had perforation of tympanic membrane
* The perforations are all dry at the time of surgery and have been dry for at least 3 months.
* No contraindication for local or general anesthesia.
* No recent upper respiratory tract infection at least 2 weeks before surgery.
* No unstable underlying condition.
* Have at least 2 months of follow up.
* Agree to participate in the study
* Aaccept to be randomized to receive treatment
* Willing to sign an informed consent

Exclusion Criteria:

* Medial placing or inlay surgical technique
* Chronic otitis media
* Contraindication of vasoconstriction agent (adrenaline)
* Allergy to analgesic agent (Xylocaine or Lidocaine)
* Concomitant with mastoiditis.
* Previous intracranial or extra-cranial complication of chronic otitis media.
* Pregnancy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score, evaluated by Visual analogue scale. | 24 hour postoperative.
  Evaluate pain score by Visual analogue scale. Patients are asked to score their pain on visual analogue scale at 4 hour, 24 hour and 48 hour postoperative.

SECONDARY OUTCOMES:
Audiometric parameters | 20th week postoperative
  Evaluated by audiometry (pure tone average of air and bone conduction, air-bone gap.)
The intactness of graft, evaluated by endoscopic visualization, and is catergorized as perforated or healed. | 20th week postoperative.
  The intactness of graft is evaluated by endoscopic visualization, and is catergorized as perforated or healed.
Operative time | Begining to the end of surgery
  The actual operating time is recorded from beginning of local anesthetic injection to the end of the surgery (complete skin suturing).

CONTACTS AND LOCATIONS:
Overall Officials: Yuvatiya Plodpai, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand